CLINICAL TRIAL: NCT03380364
Title: Role of Routine Hysteroscopy in Management of Cases of Unexplained Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Habib, dr, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: routine hysteroscopy
Record Dates: First submitted 2017-12-17; First posted 2017-12-21 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Unexplained Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Undergoing Hysterosopy (Experimental): This group will include 75 women with unexplained infertility. 5 mm rigid sheath Office hysteroscopy will be performed during the proliferative phaseof the menstrual cycle.
  Interventions: Device: hystroscope

INTERVENTIONS:
Device: hystroscope — Procedure: Hysteroscopy Office hysteroscopy will be performed during the proliferative phaseof the menstrual cycle.
  All OH (office hysteroscopy) procedures will be performed with a vaginoscopic approach without utilizing a speculum and applying traction to the cervix with a tenaculum.
  Antibiotic prophylaxis: None OH will be cancelled until after treatment of vaginal infection.
  Other Name: ROH: Routine Office Hysteroscopy Device: Hysteroscope The device used is a rigid hysteroscope (continuous flow, 30 degree forward oblique view) assembled in a 5-mm diameter diagnostic rigid sheath with an atraumatic tip (Karl Storz Endoscopy).
  Illumination: High intensity cold light source and fiberoptic cable Distention medium: solution of 0.9% normal saline with pressure at 100-120 mmHg

SUMMARY:
The aim of this work is to assess the value of hysteroscopy in unexplained infertility.

DETAILED DESCRIPTION:
The diagnosis of unexplained infertility is one of exclusion and is made only after an infertility evaluation has failed to reveal abnormalities. There is no consensus on which tests should be performed before making this diagnosis (Salim et al., 2011).

The Europe society for human and embryology (ESHRE) suggested standard diagnostic tests for infertility evaluation. These tests include semen analysis, demonstration of tubal patency by hystosalpingography (HSG) or laparascopy and laboratory assessment of ovulation (Polisseni et al., 2003). Moreover post coital test has been included by some authors as a fundamental requirement before the diagnosis of unexplained infertility while other authors found that it is unnecessary however conducting additional investigation and treating any abnormalities detected may be effective in management of women with unexplained infertility especially in older couples (Wortman et al., 2013).

For evaluation of the uterine cavity, the basic work-up consists of transvaginal sonography (TVS) with or without the use of saline or gel as a contrast medium, possibly followed by either HSG or hysteroscopy to directly assess the uterine cavity.

Both TVS, as well as saline infusion sonography (SIS) and gel instillation sonography (GIS) are inexpensive, non-invasive and have been shown to be excellent diagnostic tool to detect subtle intrauterine abnormalities (Rodrigues et al., 2014).

However, hysteroscopy allows direct visualization of the endometrial lining and detects multiple lesions and subtle uterine abnormalities that cannot be identified by the previous techniques. Moreover, hysteroscopy enables treatment of small uterine pathology in the same setting. Therefore, it is frequently referred to as the golden standard. Many studies have concluded that whenever laparoscopy is performed, it should be combined with hysteroscopy in order to complete the assessment before starting the infertility treatment (Chan et al., 2011).

In the assisted reproductive technique, a number of studies was conducted on women before in vitro fertilization (IVF) cycle revealed that the prevalence of un suspected intra uterine abnormalities, diagnosed by hysteroscopy prior to IVF cycles was 11% - 45% (Shokeir et al., 2011).

Although the role of these subtle lesions as a cause of infertility is debatable,( Kilic et al., 2013) hysteroscopic assessment and treatment of any abnormalities detected has improved the clinical pregnancy rate , live birth, and considered cost effective before IVF cycles (Grimbizis et al., 2003) .

It is widely accepted that a complete infertility workup includes an evaluation of the uterine cavity (Chan et al., 2011). Uterine abnormalities, congenital or acquired, are implicated as one of the causes of infertility. In fact, infertility related to uterine cavity abnormalities has been estimated to be the causal factor in as many as 10% to 15% of couples seeking treatment (Romani et al. 2013).

Hysteroscopy enables visualisation of the uterine cavity and allows the diagnosis and surgical treatment of intrauterine pathology. (Umranikar et al., 2016). Direct view of uterine cavity offers a significant advantage over other blind or indirect diagnostic methods. Although , hystrosalpingography (HSG) is reported to be as accurate as hysteroscopy in the diagnosis of normal and abnormal cavities, the nature of intrauterine filling defects is more accurately revealed by hysteroscopy (Jenneke et al.,2013).

The role of hysteroscopy in infertility investigation is to detect possible intrauterine change that could interfere with implantation or growth, or both, of the conceptus (Scholten et al., 2013) and to evaluate the benefit of direct treatment modalities in restoring a normal endometrial environment (Prasanta et al., 2013).

Several studies have been also performed to find out that if hystroscopic treatment of intrauterine pathologies increases the cause of failure of IVF-ET (Fatemi et al., 2010) and therefore hysteroscopy should be a part of infertility workup for all patients prior to undergoing IVF treatment and have also recommended screening of the uterus by hysteroscopy before proceeding with IVF/ICSI, to minimize implantation failure (Ryan et al. 2005).

The potential risk of diagnostic hysteroscopy are rare in most series (0-1%) especially in office procedure (John et al., 2013), while (5-24%) of operative cessions may result in intraoperative or early postoperative complications which include infection, bleeding, and even perforation of the uterus. Certain factors are considered contraindication to hystroscope like PID (Aydeniz et al., 2004).

ELIGIBILITY:
Inclusion Criteria:

* 1. All women aged (20-35) years old. 2. Unexplained infertility

Exclusion Criteria:

* 1. Female genital tract cancer, including cervical or uterine cancer 2. Active pelvic infection 3. Known uterine factor for infertility.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 6 months
  Biochemical and clinical Pregnancy Biochemical pregnancy will be determined by a positive pregnancy test performed 1week after a missed period and clinical pregnancy will be defined by the presence of a gestational sac using transvaginal ultrasound performed 6 weeks after a missed period.

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Al helaly, PhD, Study Director — Ain Shams University (Obs&Gyn); Kaled S Mohamed, PhD, Study Chair — Ain Shams University (Obs&Gyn)
Locations (1):
- Department of obstetrics and gynaecology, faculty of medicine, Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aydeniz B, Gruber IV, Schauf B, Kurek R, Meyer A, Wallwiener D. A multicenter survey of complications associated with 21,676 operative hysteroscopies. Eur J Obstet Gynecol Reprod Biol. 2002 Sep 10;104(2):160-4. doi: 10.1016/s0301-2115(02)00106-9. PMID 12206931
- [Result] Chan YY, Jayaprakasan K, Zamora J, Thornton JG, Raine-Fenning N, Coomarasamy A. The prevalence of congenital uterine anomalies in unselected and high-risk populations: a systematic review. Hum Reprod Update. 2011 Nov-Dec;17(6):761-71. doi: 10.1093/humupd/dmr028. Epub 2011 Jun 24. PMID 21705770
- [Result] Chan YY, Jayaprakasan K, Tan A, Thornton JG, Coomarasamy A, Raine-Fenning NJ. Reproductive outcomes in women with congenital uterine anomalies: a systematic review. Ultrasound Obstet Gynecol. 2011 Oct;38(4):371-82. doi: 10.1002/uog.10056. PMID 21830244
- [Result] Fatemi HM, Kasius JC, Timmermans A, van Disseldorp J, Fauser BC, Devroey P, Broekmans FJ. Prevalence of unsuspected uterine cavity abnormalities diagnosed by office hysteroscopy prior to in vitro fertilization. Hum Reprod. 2010 Aug;25(8):1959-65. doi: 10.1093/humrep/deq150. Epub 2010 Jun 22. PMID 20570971
- [Result] Grimbizis GF, Camus M, Tarlatzis BC, Bontis JN, Devroey P. Clinical implications of uterine malformations and hysteroscopic treatment results. Hum Reprod Update. 2001 Mar-Apr;7(2):161-74. doi: 10.1093/humupd/7.2.161. PMID 11284660
- [Result] Kasius JC, Eijkemans RJ, Mol BW, Fauser BC, Fatemi HM, Broekmans FJ. Cost-effectiveness of hysteroscopy screening for infertile women. Reprod Biomed Online. 2013 Jun;26(6):619-26. doi: 10.1016/j.rbmo.2013.02.015. Epub 2013 Mar 14. PMID 23602685
- [Result] Keats JP. Patient safety in the obstetric and gynecologic office setting. Obstet Gynecol Clin North Am. 2013 Dec;40(4):611-23. doi: 10.1016/j.ogc.2013.08.004. PMID 24286992
- [Result] Kilic Y, Bastu E, Ergun B. Validity and efficacy of office hysteroscopy before in vitro fertilization treatment. Arch Gynecol Obstet. 2013 Mar;287(3):577-81. doi: 10.1007/s00404-012-2584-z. Epub 2012 Oct 6. PMID 23053317
- [Result] Polisseni F, Bambirra EA, Camargos AF. Detection of chronic endometritis by diagnostic hysteroscopy in asymptomatic infertile patients. Gynecol Obstet Invest. 2003;55(4):205-10. doi: 10.1159/000072075. PMID 12904693
- [Result] Nayak PK, Mahapatra PC, Mallick J, Swain S, Mitra S, Sahoo J. Role of diagnostic hystero-laparoscopy in the evaluation of infertility: A retrospective study of 300 patients. J Hum Reprod Sci. 2013 Jan;6(1):32-4. doi: 10.4103/0974-1208.112378. PMID 23869148
- [Result] Ray A, Shah A, Gudi A, Homburg R. Unexplained infertility: an update and review of practice. Reprod Biomed Online. 2012 Jun;24(6):591-602. doi: 10.1016/j.rbmo.2012.02.021. Epub 2012 Mar 7. PMID 22503948
- [Result] Romani F, Guido M, Morciano A, Martinez D, Gaglione R, Lanzone A, Selvaggi L. The use of different size-hysteroscope in office hysteroscopy: our experience. Arch Gynecol Obstet. 2013 Dec;288(6):1355-9. doi: 10.1007/s00404-013-2932-7. Epub 2013 Jun 25. PMID 23797933
- [Result] Ryan GL, Syrop CH, Van Voorhis BJ. Role, epidemiology, and natural history of benign uterine mass lesions. Clin Obstet Gynecol. 2005 Jun;48(2):312-24. doi: 10.1097/01.grf.0000159538.27221.8c. No abstract available. PMID 15805789
- [Result] Salim S, Won H, Nesbitt-Hawes E, Campbell N, Abbott J. Diagnosis and management of endometrial polyps: a critical review of the literature. J Minim Invasive Gynecol. 2011 Sep-Oct;18(5):569-81. doi: 10.1016/j.jmig.2011.05.018. Epub 2011 Jul 23. PMID 21783430
- [Result] Scholten I, Moolenaar LM, Gianotten J, van der Veen F, Hompes PG, Mol BW, Steures P. Long term outcome in subfertile couples with isolated cervical factor. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):429-33. doi: 10.1016/j.ejogrb.2013.06.042. Epub 2013 Aug 3. PMID 23921361
- [Result] Shokeir T, Abdelshaheed M, El-Shafie M, Sherif L, Badawy A. Determinants of fertility and reproductive success after hysteroscopic septoplasty for women with unexplained primary infertility: a prospective analysis of 88 cases. Eur J Obstet Gynecol Reprod Biol. 2011 Mar;155(1):54-7. doi: 10.1016/j.ejogrb.2010.11.015. Epub 2010 Dec 23. PMID 21185112
- [Result] Umranikar S, Clark TJ, Saridogan E, Miligkos D, Arambage K, Torbe E, Campo R, Di Spiezio Sardo A, Tanos V, Grimbizis G; British Society for Gynaecological Endoscopy /European Society for Gynaecological Endoscopy Guideline Development Group for Management of Fluid Distension Media in Operative Hysteroscopy. BSGE/ESGE guideline on management of fluid distension media in operative hysteroscopy. Gynecol Surg. 2016;13(4):289-303. doi: 10.1007/s10397-016-0983-z. Epub 2016 Oct 6. No abstract available. PMID 28003797
- [Result] Wortman M, Daggett A, Ball C. Operative hysteroscopy in an office-based surgical setting: review of patient safety and satisfaction in 414 cases. J Minim Invasive Gynecol. 2013 Jan-Feb;20(1):56-63. doi: 10.1016/j.jmig.2012.08.778. Epub 2012 Oct 27. PMID 23107759